CLINICAL TRIAL: NCT06257901
Title: Co-design of a Physical Activity and Sedentary Behaviour Intervention for Adults with Fabry Disease
Brief Title: A Co-designed Physical Activity Intervention in Fabry Disease
Status: Completed | Type: Observational
Sponsor: Brunel University (Other)
Collaborators: Royal Free Hospital NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr Daniel Bailey, Senior Lecturer in Sport, Health and Exercise Sciences, Brunel University
Other Study IDs: 45091-NHS-Oct/2023- 47368-1
Record Dates: First submitted 2024-01-25; First posted 2024-02-14 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Adults with Fabry disease: Focus groups and participatory workshops
  Interventions: Other: Interviews/Focus groups/Participatory workshops
- Lay specialist stakeholders: Focus groups
  Interventions: Other: Interviews/Focus groups/Participatory workshops
- Specialist stakeholders: Interviews
  Interventions: Other: Interviews/Focus groups/Participatory workshops

INTERVENTIONS:
Other: Interviews/Focus groups/Participatory workshops — Qualitative study (no intervention delivered)

SUMMARY:
Currently, treatments for Fabry disease are pharmacological and predominantly focus on the physical symptoms of the disease. In the general population and individuals with disabilities, increasing physical activity levels and reducing sedentary time can be an effective, non-pharmacological treatment to improve mental health and quality of life. Such interventions have not yet been developed or evaluated in people with Fabry disease.

The aim of this study is to co-design a physical activity and sedentary behaviour intervention tailored to the needs of adults with Fabry disease. The study will seek to gain the expertise of adults with Fabry disease, specialist stakeholders (physicians, cardiologists and clinical nurse specialists) and lay specialist stakeholders (family and friends of adults with Fabry disease and members of staff and volunteers at the Society for Mucopolysaccharide Diseases). A range of views and experiences of physical activity and sedentary behaviour will be explored via focus groups (with individuals with Fabry disease and lay specialist stakeholders) and semi-structured interviews (with specialist stakeholders). The information gathered from the focus groups and interviews will then be utilised to inform participatory workshops (with individuals with Fabry disease) to test intervention concepts. Data from these activities will inform the design of a future intervention.

ELIGIBILITY:
Individuals with Fabry disease will be eligible to participate in the study if they meet the following inclusion criteria:

* Have been diagnosed with Fabry disease.
* Aged ≥ 18 years old.
* Able to independently ambulate with or without the use of a walking aid.
* Lives in the United Kingdom.
* Deemed eligible to participate following screening by a clinician (for participatory workshops).

The circumstances in which an individual may be deemed ineligible to participate in the participatory workshops based on the clinician's assessment are as follows:

* Severe neuropathic pain.
* Stage 4 heart failure or other condition resulting in breathlessness to a level they cannot participate.
* Other clinical condition which dominates the clinical picture to the extent that it dominates the symptoms and biases the results.

Exclusion criteria for all participants will be as follows:

* Incapacity to provide written informed consent.
* Unable to communicate in English to a sufficient level to permit engagement in the study.

Specialist stakeholders will be members of staff at NHS specialist centres for Fabry disease who are directly involved in the healthcare of adults with Fabry disease.

Lay specialist stakeholders will be individuals who have been involved in supporting adults with Fabry disease, such as family, friends and members of staff at the Society for Mucopolysaccharide Diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adults with Fabry disease, lay specialist stakeholders and specialist stakeholders who meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 41 (Actual)
Dates: Start 2024-03-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Focus groups (adults with Fabry disease) | 9 months
  Themes describing adults with Fabry disease's views and experiences of physical activity and sedentary behaviour- Emergence of themes describing participants' views and experiences from analysis of focus groups (using the Framework Method).
Focus groups (lay specialist stakeholders) | 9 months
  Themes describing lay specialist stakeholders' views and experiences of physical activity and sedentary behaviour- Emergence of themes describing participants' views and experiences from analysis of focus groups (using the Framework Method).
Semi-structured interviews (specialist stakeholders) | 9 months
  Themes describing specialist stakeholders' views and experiences of physical activity and sedentary behaviour- Emergence of themes describing participants' views and experiences from analysis of interviews (using the Framework Method).
Participatory workshops (adults with Fabry disease) | 9 months
  Themes describing adults with Fabry disease's views and experiences of initial intervention concepts- Emergence of themes describing participants' views and experiences from analysis of participatory workshops (using the Framework Method).

CONTACTS AND LOCATIONS:
Locations (1):
- Brunel University London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No